CLINICAL TRIAL: NCT00966407
Title: Assessing Inherited Markers of Metabolic Syndrome in the Young
Acronym: AIMMY
Status: Completed | Type: Observational
Sponsor: Eric Hoffman (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Howard University (Other); University of Massachusetts, Worcester (Other); East Carolina University (Other)
Responsible Party: Sponsor-Investigator, Eric Hoffman, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: CNMC IRB#3842; 2P20MD000198-06 (NIH)
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Metabolic Syndrome; Diabetes Mellitus, Type 2; Obesity
Keywords: Metabolic Syndrome; Obesity; Genetic risk markers; Single Nucleotide Polymorphisms; Young adults; Fitness testing
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples are obtained for DNA extraction and measuring various biomarkers (including fasting glucose, insulin, lipid profile, and hemoglobin A1c)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Young Adults: College-age (18-35 years) participants recruited from Howard University, East Carolina University, and University of Massachusetts, Amherst, University of Calgary, Winston-Salem University

SUMMARY:
The AIMM Young study is a collaboration between Children's National Medical Center (CNMC) and colleges/universities nationwide--currently including Howard University (HU), East Carolina University (ECU), and University of Massachusetts, Amherst (U Mass). This study obtains a variety of baseline measures (such as serum biomarkers related to metabolic syndrome, anthropometrics, muscle strength, and fitness testing) along with genetic information from healthy college-age (18-35 years) young adults in efforts to identify phenotype-genotype associations that may predispose individuals to developing metabolic syndrome, type 2 diabetes, and/or related diseases such as obesity.

We hypothesized that certain genetic variations will be protective against metabolic syndrome, while others will show a strong correlation with specific components of metabolic syndrome disease. We expect that the study of "pre-symptomatic," young individuals will facilitate the identification of genetic risk loci for metabolic syndrome and type 2 diabetes. Younger populations typically have less confounding variables, and this facilitates normalizing of metabolic syndrome features and environment/lifestyle. Additionally, young subjects can provide more robust longitudinal data, and be recruited into subsequent interventions to reverse the trend towards metabolic syndrome, rather than the more difficult task of reversing type 2 diabetes in older populations. The data collected will be stratified according to gender, age, ethnicity, genotype, and other phenotypic measures to determine how these factors influence disease risk.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 35 years
* post-puberty
* willing and able to provide informed consent
* stable medical and psychosocial status providing a high likelihood of follow-up and compliance with study protocol
* all ethnic backgrounds will be included in this study.

Exclusion Criteria:

* evidence of clinically relevant systemic disease associated with disorders of glucose metabolism
* chronic use of glucocorticoid or appetite suppressants
* concomitant use of drugs known to alter glucose metabolism (i.e., metformin, thiazolidinediones, sulfonylurea receptor agonists and inhibitors of alpha-glucoside hydrolase) or other medications known to alter blood levels being tested in this study
* inability to provide the requested fasting blood sample
* pregnancy
* menopause
* alcohol dependency (as determined by CAGE screening questionnaire); (8) inability to provide informed consent
* previous diagnosis or treatment for any hematologic-oncologic disorder
* history or current treatment for an eating disorder
* current treatment for weight loss
* history of bariatric surgery
* history of neurosurgical procedure
* participation in another clinical trial involving an investigational drug
* history of psychiatric disorder, which in the opinion of the investigator would affect the conduct of the proposed trial
* age younger than 18 or older than 35 at the time of recruitment
* weight that exceeds the capacity of equipment used for weight measurements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population from which cohorts will be selected include students, residents, staff, and/or faculty who are present on Howard University, East Carolina University, and/or University of Massachusetts, Amherst campuses and surrounding areas.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Genotype for specific genes related to obesity, metabolic syndrome, and/or type 2 diabetes; Fasting serum biomarkers; Hand grip strength, muscle strength of upper and lower extremities; Fitness measurements; Body composition measures | Cross-sectional, one-time measure

SECONDARY OUTCOMES:
Perception of physical fitness; Relationship between physiological measures and genotype variation | Cross-sectional, one-time

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Hoffman, Ph.D, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Deschamps CL, Connors KE, Klein MS, Johnsen VL, Shearer J, Vogel HJ, Devaney JM, Gordish-Dressman H, Many GM, Barfield W, Hoffman EP, Kraus WE, Hittel DS. The ACTN3 R577X Polymorphism Is Associated with Cardiometabolic Fitness in Healthy Young Adults. PLoS One. 2015 Jun 24;10(6):e0130644. doi: 10.1371/journal.pone.0130644. eCollection 2015. PMID 26107372
- [Result] Many GM, Lutsch A, Connors KE, Shearer J, Brown HC, Ash G, Pescatello LS, Gordish-Dressman H, Barfield W, Dubis G, Houmard JA, Hoffman EP, Hittel DS. Examination of Lifestyle Behaviors and Cardiometabolic Risk Factors in University Students Enrolled in Kinesiology Degree Programs. J Strength Cond Res. 2016 Apr;30(4):1137-46. doi: 10.1519/JSC.0000000000000871. PMID 25647655
- [Result] Karlos A, Shearer J, Gnatiuk E, Onyewu C, Many G, Hoffman EP, Hittel DS. Effect of the SORT1 low-density lipoprotein cholesterol locus is sex-specific in a fit, Canadian young-adult population. Appl Physiol Nutr Metab. 2013 Feb;38(2):188-93. doi: 10.1139/apnm-2012-0231. Epub 2012 Nov 1. PMID 23438231
- [Result] Arnold TJ, Schweitzer A, Hoffman HJ, Onyewu C, Hurtado ME, Hoffman EP, Klein CJ. Neck and waist circumference biomarkers of cardiovascular risk in a cohort of predominantly African-American college students: a preliminary study. J Acad Nutr Diet. 2014 Jan;114(1):107-16. doi: 10.1016/j.jand.2013.07.005. Epub 2013 Sep 16. PMID 24051106